CLINICAL TRIAL: NCT00651248
Title: Evaluation of Salivary Flow and Buffer Capacity Associated to Aged People's Oral Health
Status: Completed | Type: Observational
Sponsor: Academia Cearense de Odontologia (Other)
Responsible Party: Maria Vieira de Lima Saintrain, Universidade de Fortaleza
Other Study IDs: renatago
Record Dates: First submitted 2008-03-31; First posted 2008-04-02 (Estimated); Last update posted 2008-04-02 (Estimated); Status verified 2008-03

CONDITIONS: Oral Health; Diagnosis, Oral; Public Health
Keywords: Saliva; Oral health; Aged
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to identify the relation of the salivary flow and the buffer capacity of the saliva with medicine, buccal discomfort and auto-related illnesses in aged people.

DETAILED DESCRIPTION:
Study clinical of prevalence. 68 aged, average 70.4 years, SD ± 7.27 represented institution's residents of long permanence. Questionnaire was applied, organizing the data for Software SPSS version 15. The test qui-square of Pearson was used, level of significance 5% and reliable interval 95%. 80% presented pH normal. The salivary Flow: 32.3% very low, 41.2% reduced and 25.5% normal. 30.9% mentioned dry mouth, 22.1% tasting's problems, 17.6% dysphagia and 14.7% burning mouth. Main systemic illnesses: 48.5% declared cardiovascular problems, 17.6% diabetes and 16.2% osteoporosis. 76.5% used medicine. There was a significance statistic between medicine taking and dry mouth (p=0.013), buffer capacity and burning mouth (p=0.019), salivary flow and medicine taking (p=0.048). The low salivary flow and the buffer capacity of the saliva influence in the aged people's health condition, as the drugs influence the results.

ELIGIBILITY:
Inclusion Criteria:

* aged people with 60 years old or more,
* ills or not,
* able to realize tests
* people who want to participate of research

Exclusion Criteria:

* people less 60 years old

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 68 aged, average 70.4 years, SD ± 7.27 represented institution's residents of long permanence.
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2006-09; Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria VL Saintrain, doutor, Principal Investigator — Universidade de Fortaleza
Locations (1):
- Instituição de Longa Permanência Lar Torres de Melo, Fortaleza, Ceará, Brazil